CLINICAL TRIAL: NCT03346421
Title: Assessment of Anthropometric Parameters, Protein and Metabolic Profile and Function of the Respiratory System in Obese Patients Reducing Their Body Mass Under Controlled Conditions
Brief Title: Anthropometric Parameters, Metabolic Profile and Function of the Respiratory System in Obese Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Agnieszka Zawada, principal investigator, Poznan University of Medical Sciences
Other Study IDs: AofMPRinO
Record Dates: First submitted 2017-10-04; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Obesity; Diet Modification; Physical Activity
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Diet; Exercise

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- diet and physical activity
  Interventions: Behavioral: diet and physical activity

INTERVENTIONS:
Behavioral: diet and physical activity

SUMMARY:
Obesity is currently considered an increasingly more severe social and health related problem. The World Health Organization qualified obesity as a chronic disease along with circulatory diseases, diabetes, cancer and respiratory diseases. The principal physiological methods of treatment for this disease are diet and exercise. The aim of the study is assess anhtropometric parameters, metabolic and proteomic profile and respiratory truck function in obese patients reducing body weight during 21 days course of calorie restriction and physical activity.

DETAILED DESCRIPTION:
THE AIM OF THE STUDY:

Determining changes in anthropometric parameters, both the protein and metabolic profile as well as changes in the respiratory system functional testing in obese patients, in whom an attempt to reduce body mass (through dietary treatment and physical activity), under controlled conditions (over a period of a 21-day hospitalization) was made.

RESEARCH METHODOLOGY:

The study will be conducted on a group of a 100 persons with obesity who fulfilled the inclusion criteria (index BMI>30 kg/m2/ and an increased adipose tissue content assessed by the electrical bioimpedance method)

RESEARCH PLAN

I. The research will include studies conducted in The Department and Clinic of Gastroenterology, Dietetics and Internal Medicine in Poznan, performed by members of the research team, before and after a 21-day weight loss cycle:

1. The assessment of anthropometric parameters (height, body mass, BMI, the waist and hip circumference, the WHR index) and the assessment of the body adipose tissue content using the electrical bioimpedance method, with TANITA MC-980 MA TANITA AB140 ViScan device).
2. The detailed medical history, considering other parameters that may influence an increase in body mass, based on a detailed specially prepared questionnaire (regarding disease history, socio-economical data and eating habits).
3. Objective and subjective assessment, systolic and diastolic blood pressure measurement (two-time measurement with the sphygmomanometer using the Korotkow method, in a sitting position, after a 5 minute rest), as well as a systolic and diastolic blood pressure measurement in reaction to verticalization.

The following parameters will be assessed in a study group:

1. Lipid parameters (the total cholesterol density, HDL fraction, LDL and the triglycerides in the serum) using the enzymatic method. The HDL cholesterol will be calculated based on the following formula: nonHDL cholesterol = total cholesterol - HDL fraction cholesterol and the ratio TG/HDL will be calculated as well.
2. Inflammatory response markers assessment, OB and CRP, using a standard method
3. Liver function assessment (ALT, AST, GGTP) using a standard method.
4. Kidney function assessment (the creatinine concentration in the serum including the estimated indicator of glomerular filtration rate (eGFR) according to the Modification of Diet Renal Disease Study Equation (MDRD) norm: 90-120ml/min/1,73 m². CChN will be classified according to the estimated indicator of glomerular filtration rate: stage G1 (eGFR≥90 ml/min/1,73 m²), stage G2 (eGFR 60-89 ml/min/1,73 m²), stage G3a (eGFR45-59 ml/min/1,73 m²), stage G3b (eGFR30-45 ml/min/1,73 m²) stage G4 (eGFR 5-29 ml/min/1,73 m²) and stage G5 (eGFR<15 ml/min/1,73 m² or dialysis treatment). [1] The plan is to assess, within the study group, the albumin/creatinine index in a morning urine sample. The value of the albumin/creatinine index>30mg/g will be considered positive.
5. The evaluation of markers: alfa-fetoprotein, Ca19,9, CEA using a standard method.

Furthermore, the patients will be asked to fill out additional questionnaires:

1. Questionnaire evaluating the eating behavior and opinion on food and nutrition (QEB) and a Physical activity questionnaire
2. Questionnaires assessing the quality of sleep: (Athens Insomnia Scale and Pittsburgh Sleep Quality Index (PSQI).
3. Sleep apnea scale
4. Psychological surveys: Multidimensional Health Locus and Control Scale (MHLC), Satisfaction with Life Scale (SWLS), Acceptance of Illness Scale (AIS)
5. Additionally for patients with accompanying diabetes: Problem Areas in Diabetes (PAID) Diabetes Treatment Questionnaire (DTSQ) II. 21-day stay in the Greater Poland Pulmonology and Thoracic Surgery Centre, The Department of Pulmonology and Rehabilitation (Unit in Ludwikowo near Poznan)

Indications for hospitalization:

1. Obesity disenabling professional work and social function performing.
2. Necessity of body mass reduction to improve lipid parameters
3. Sleep disorder caused by excess body mass (sleep apnea syndrome)
4. Pre-diabetes or diabetes related to accompanying obesity
5. Osteoarticular system disorders related to obesity disenabling the execution of planned orthopedic procedures

The following will be conducted on subjects of the study during hospitalization:

1. A 21-day body mass reduction attempt will be implemented under sanatorial conditions. A rational hypo-calorie diet will be applied to all patients (calorie reduction proportional to the BMR calculated into actual body mass, macro-elements: 15-20% protein, 25-30% fat, 50-55% carbohydrates, simple sugar content <5%, dietary fiber 30g)
2. Throughout a period of the weight loss program the following will be implemented: standard motor rehabilitation - kinesitherapy (2 x a day for 25 minutes), stationary bike training (1x a day for 10 minutes) as well as passive mechanical exercises (1x a day for 15 minutes), abdominal muscle exercises (1x a day with an increasing, by 10, number of repetitions starting with 30).
3. Every patient will also take two physiotherapeutic treatments recommended by a physiotherapist (laser, ultrasounds, TENS, magnetic field, iontophoresis).
4. The following respiratory system tests will be conducted before the beginning as well as on the 21-st day of the weight loss cycle: arterial blood gasometry, spirometry, ergospirometry, body plethysmography, diffusing capacity of the lung for carbon dioxide (DLCO).
5. Furthermore, on the starting day of the program as well as after 21 days, the measurement of neck circumference and neck adipose tissue will be performed.
6. Each patient, who will be taking part in the study, will be educated in the aspect of correct nutrition and rational reduction diet rules (3 meetings -30 minutes each, conducted at 7 day intervals).
7. Furthermore, the oxidative stress parameters and the inflammatory response markers will be evaluated both at the beginning and at the end of the hospitalization period.

III. The assessment of amino acid concentration and the metabolic profile evaluation will be performed in the Department of Inorganic and Analytical Chemistry.

1. Evaluation of the protein profile will be performed using the mass spectrometer MALDI ToF/ToF,
2. The serous amino acid concentration will be performed using the mass spectrometer QTRAP 4000)
3. The Biocrates AbsolutelDQ p180 Kit will be used to evaluate the metabolic panel (glycerolophospholipids, sphingolipids).
4. Venous blood, in the amount of 20 ml will be used in order to assess parameters listed above. Determination of the above parameters will be performed twice, before and after the end of each stage (40 ml of venous blood will be sampled from each patient throughout the duration of the study).

IV. The evaluation of hormones released by the muscle and adipose tissue, the concentration of free oxygen radicals, and the total oxidation capacity in plasma will be assessed from blood samples obtained at the beginning and at the end of the 21 day study period in The Academy of Physical Education The Department of Physiology.

ELIGIBILITY:
Inclusion Criteria:

1. patient's age: above 18 years of age
2. BMI obesity >30kg/m2
3. increased content of overall adipose tissue measured by bioelectrical impendance method
4. consent to take part in the study

Exclusion Criteria:

1. positive electrocardiographic stress test
2. staying on a vegetarian or any other alternative diet
3. patients with active or post cancerous disease (ongoing radiation-/chemotherapy treatment),
4. patients with liver diseases (ALT > 3x border line ) except for patients with fatty live disease,
5. chronic kidney disease eGFR <30 ml/ 1,73m2 / min,
6. acute inflammation CRP > 5mg/dl,
7. unstable ischeamic heart disease, state after bypass surgery, implanted heart stimulator- (cardioverter, defibrillator - ICD, heart pacemaker), endovascular prosthesis,
8. patients after an ischemic or haemorrhagic stroke (<6 months)
9. post STEMI patients with a drug-eluting stent implantation, nSTEMI (<12 months)
10. inherited metabolic disorders: phenylketonouria, galactosaemia
11. autoimmune diseases (an acute thyroiditis, celiac disease, systemic connective tissue disease, haemolytic anemia, vitiligo, addison's disease, hyperbilirubinemia),
12. non specific enteneritis (Crohn's disease, ulcerative colonitis)
13. pregnancy,
14. psychological disorders, eating disorders such as anorexia, bulimia,
15. antibiotic therapy, steroid therapy, (ongoing)
16. drug, alcohol addiction (a daily consumption of more then 1 portion of alcohol).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted on a group of a 100 persons with obesity who fulfilled the inclusion criteria (index BMI>30 kg/m2/ and an increased adipose tissue content assessed by the electrical bioimpedance method).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-02-01 (Actual); Primary Completion 2018-12-21 (Estimated); Study Completion 2020-12-21 (Estimated)

PRIMARY OUTCOMES:
adipose tissue | after 12 months
  The assessment of the body adipose tissue content using the electrical bioimpedance device- TANITA MC-980 MA.( Percentage )
Satisfaction with Life Scale | after 12 months
  SWLS Questionaire
Respiratory system tests | after 12 months
  spirometry (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poland